CLINICAL TRIAL: NCT02981394
Title: Clinical Outcomes of Autologous Bone Marrow Aspirate Concentrate Injections for Musculoskeletal Conditions
Status: Withdrawn | Type: Observational
Why Stopped: No active enrollment of patients.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16090710-IRB01
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Musculoskeletal Pain; Osteoarthritis; Tendinopathy; Sprains Strain
MeSH Terms: conditions — Musculoskeletal Pain; Osteoarthritis; Tendinopathy; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (1):
- BMAC Group: Intervention Group
  Interventions: Procedure: Bone Marrow Aspirate Concentrate Injection

INTERVENTIONS:
Procedure: Bone Marrow Aspirate Concentrate Injection — BMAC will be collected in the outpatient setting with local anesthesia. The collection site will be the Posterior Superior Iliac Spine (PSIS). This will be visualized under ultrasound prior to collection. Local anesthesia with 1% lidocaine will be performed prior to the harvest. BMAC harvest will be performed using the Arthrex Angel BMAC System using the Arthrex collection protocol. The Arthrex Angel machine will be used to separate BMAC contents for injection based on Arthrex collection protocol. Machine settings, volume of collection and volume of output have not been standardized and will be based upon harvest and the condition treated. These will be variables recorded for consideration of optimal settings based on the patient-reported outcomes.

SUMMARY:
The use of Bone Marrow Autologous Collection (BMAC) in musculoskeletal conditions including osteoarthritis and tendon injuries has been growing. Outcome evidence continues to be sparse. The purpose of this study is collect a longitudinal case series of patient reported outcomes following BMAC injections for musculoskeletal conditions including osteoarthritis, tendinopathy and injuries to ligaments, tendons and muscles.

ELIGIBILITY:
Inclusion Criteria:

* Musculoskeletal Condition that is able to undergo an injection
* Patient requests the procedure and enrolls with agreement to pay for the procedure

Exclusion Criteria:

* Active Cancer
* Allergies to local anesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a musculoskeletal condition amenable to BMAC or PRP treatment will be enrolled upon registration for the selected procedure. Proper counseling regarding the selected procedure and alternatives will be done prior to enrollment. Patients with contraindications for the procedure will not undergo the procedure and therefore will not be enrolled. The study will be non-randomized; therefore, patient selection will be based upon patient request for the procedure after proper counseling. Counseling regarding cost of each procedure will also be provided. All costs for the procedure will be the responsibility of the patient. Proper documentation will also be signed by the patient indicating that procedure is elective and PRP/BMAC injections will not be billed to their insurance carriers. Upon enrollment, patients will be consented for the procedure and longitudinal data collection.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
WOMAC Score | 5 years
  Pain and Function Score

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Orthopeadics at Rush, Chicago, Illinois, United States